CLINICAL TRIAL: NCT07190079
Title: A Multicenter Comparative Study of Saline Contrast Electrical Impedance Tomography Method Versus CTPA in the Diagnosis of Acute Pulmonary Embolism
Brief Title: Saline Contrast Electrical Impedance Tomography Method for Diagnosis of Acute Pulmonary Embolism
Acronym: ECTPED
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ECTPED
Record Dates: First submitted 2025-09-14; First posted 2025-09-24 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Acute Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients clinically suspected with acute PE: This study will enroll adult patients (>18 years) with clinically suspected or confirmed acute pulmonary embolism (PE) presenting with acute respiratory failure, who either undergo computed tomography pulmonary angiography (CTPA) within 24 hours or are scheduled for CTPA within the next 24 hours. Eligible participants need to have an indwelling central venous catheter (internal jugular or subclavian vein) or a peripheral forearm venous line, with no restrictions on gender.
  Interventions: Diagnostic Test: Saline contrast Electrical Impedance Tomography method; Diagnostic Test: Computed Tomography Pulmonary Angiography (CTPA)

INTERVENTIONS:
Diagnostic Test: Saline contrast Electrical Impedance Tomography method — This study will enroll patients with clinically suspected or confirmed acute pulmonary embolism (PE) presenting with acute respiratory failure, who undergo electrical impedance tomography (EIT) with saline contrast within 24 hours before or after computed tomography pulmonary angiography (CTPA). The EIT procedure is performed as follows:
  1. Breath-Hold Maneuver: (1)Spontaneous breathing patients: Supine position, instructed to hold expiration for ≥8 seconds. (2)Mechanically ventilated patients: Expiratory hold (>8 sec) achieved via ventilator; deeper sedation will be applied when feasible to prolong breath-hold.
  2. Venous Access: (1)Preferred: Central venous catheter (internal jugular or subclavian vein).(2)Alternative: Peripheral forearm vein (preferably the median cubital vein).
  3. Contrast Administration:(1)Central venous route: 10 mL of 10% NaCl.(2)Peripheral venous route: 15 mL of 5% NaHCO₃.
Diagnostic Test: Computed Tomography Pulmonary Angiography (CTPA) — Patients who meet the inclusion criteria will undergo CTPA examination using conventional clinical diagnostic methods.

SUMMARY:
The goal of this observational study is to compare the consistency of saline contrast Electrical Impedance Tomography(EIT) method and Computed Tomography Pulmonary Angiography (CTPA) in diagnosing acute pulmonary embolism. The main question it aims to answer is:

Can bedside saline contrast EIT method be used for the diagnosis of acute pulmonary embolism? The participants will undergo saline contrast EIT and CTPA examinations successively within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinically suspected or confirmed acute pulmonary embolism (PE) presenting with acute respiratory failure;
2. Availability of CTPA results within 24 hours or scheduled to undergo CTPA within the next 24 hours;
3. Age >18 years; no gender restrictions;
4. Presence of central venous access (internal jugular or subclavian vein) or peripheral forearm venous access;
5. Willingness to participate with signed informed consent from either the patient or legal guardian.

Exclusion Criteria:

1. Pregnancy or lactation;
2. Relative contraindications to EIT examination (e.g., chest wall wounds at electrode belt placement site, presence of pacemakers);
3. Severe hypernatremia (serum sodium >155 mmol/L);
4. Inability to maintain expiratory breath-hold for ≥8 seconds;
5. BMI >50 or severe thoracic deformities;
6. Current extracorporeal membrane oxygenation (ECMO) therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinically suspected or confirmed acute pulmonary embolism (PE) presenting with acute respiratory failure.
Sampling Method: Non-Probability Sample
Enrollment: 343 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
The ability of proportion of dead space ventilation to diagnose PE | Within 24 hours before or after the CTPA examination
  The participant undergoes a saline contrast EIT examination, after which the distribution of pulmonary ventilation and perfusion will be obtained, respectively. A V-Q map will be subsequently generated. Using offline EIT data analysis tool, the proportion of lung regions with ventilation but without perfusion is calculated, representing the proportion of dead space ventilation (expressed as a percentage). Area under the receiver operating characteristic curve (AUROC), sensitivity, specificity, Youden's index, accuracy, Kappa statistic, positive predictive value (PPV), negative predictive value (NPV), positive likelihood ratio (PLR) and negative likelihood ratio (NLR) will be used to evaluate the ability of proportion of dead space ventilation to diagnose acute pulmonary embolism (PE).

SECONDARY OUTCOMES:
The ability of proportion of V/Q matching to diagnose PE | Within 24 hours before or after the CTPA examination
  Following a saline contrast EIT examination, the participant's pulmonary ventilation and perfusion distributions will be obtained, allowing for the generation of a V-Q map. Using offline EIT data analysis tool, the proportion of lung regions demonstrating both ventilation and perfusion will be calculated, representing the proportion of V/Q matching (%). Area under the receiver operating characteristic curve (AUROC), sensitivity, specificity, Youden's index, accuracy, Kappa statistic, positive predictive value (PPV), negative predictive value (NPV), positive likelihood ratio (PLR) and negative likelihood ratio (NLR) will be used to evaluate the ability of proportion of V/Q matching to diagnose acute pulmonary embolism (PE).
The ability of proportion of shunt to diagnose PE | Within 24 hours before or after the CTPA examination
  Following a saline contrast EIT examination, the participant's pulmonary ventilation and perfusion distributions will be obtained, enabling the generation of a V-Q map. Using offline EIT data analysis tool, the proportion of lung regions exhibiting perfusion without ventilation will be calculated, representing the proportion of shunt (%). Area under the receiver operating characteristic curve (AUROC), sensitivity, specificity, Youden's index, accuracy, Kappa statistic, positive predictive value (PPV), negative predictive value (NPV), positive likelihood ratio (PLR) and negative likelihood ratio (NLR) will be used to evaluate the ability of proportion of shunt to diagnose acute pulmonary embolism (PE).
The ability of other indicators reflecting pulmonary ventilation and perfusion to diagnose PE | Within 24 hours before or after the CTPA examination
  Following a saline contrast EIT examination, the participant's pulmonary ventilation and perfusion distributions will be obtained, and a V-Q map will be subsequently generated. Using offline EIT data analysis tool, additional indices reflecting pulmonary ventilation and perfusion will be further calculated. Area under the receiver operating characteristic curve (AUROC), sensitivity, specificity, Youden's index, accuracy, Kappa statistic, positive predictive value (PPV), negative predictive value (NPV), positive likelihood ratio (PLR) and negative likelihood ratio (NLR) will be used to evaluate the ability of other indicators reflecting pulmonary ventilation and perfusion to diagnose acute pulmonary embolism (PE).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care Medicine, Peking Union Medical College Hospital, Peking Union Medical College, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No